CLINICAL TRIAL: NCT05958186
Title: A Study of Cytomegalovirus Disease Epidemiology in Pediatric and Adult Liver Transplant Recipients in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Lin Zhong (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Lin Zhong, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: SHLTQC-6
Record Dates: First submitted 2023-07-12; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Cytomegalovirus (CMV) Infections Among Children and Adult Liver Transplantation Patients in China
Keywords: Cytomegalovirus; Children; Adult; Liver transplantation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and serum of recipients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children group: Ages≤18
- Adults group: Ages>18

SUMMARY:
The goal of this observational study is to learn about cytomegalovirus disease epidemiology in pediatric and adult liver transplant recipients in China. The main questions it aims to answer are:

* The incidence of Cytomegalovirus (CMV) Infections (including clinical significant CMV reactivations and CMV Diseases) among children and adults Liver transplantation patients in China
* All-cause Mortality (Survival probability at 1 year)
* Incidence of Allograft Rejection. Number of subjects with allograft rejection
* Graft Loss. Incidence of graft loss (re-transplantation)
* Late-onset CMV Disease. Incidence of late-onset CMV disease (occurring after 100 days post-randomization) as adjudicated by end point committee
* Bacterial Infections. Incidence of bacterial opportunistic infections
* Major Fungal Infections. Opportunistic fungal infections
* Major Non-CMV Viral Infections. Incidence of non-CMV viral infections We will collect demographic data of participants. All recipients and donors underwent preoperative testing for CMV pp65 antigenemia, plasma CMV DNA, and serum CMV antibody. All the recipients were followed up in a liver transplant follow-up clinic twice weekly for a month after discharge from hospital. After that, patients were followed up weekly for 3 months, fortnightly for 6 months, and monthly for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Have received their first orthotopic liver transplant (the transplanted liver may be deceased donor or live donor graft) within 10 days prior.
* Children group: Age ≤18yeas；
* Adults group: Age >18yeas；
* Willingness to participate in the study
* Ability to understand information material
* Written informed consent

Exclusion Criteria:

* Have known Human immunodeficiency virus (HIV) infection (based on testing performed during the transplant evaluation process).
* Participation in another investigational agent trial
* Be undergoing multi organ transplant or have undergone prior organ transplant. Have expected life expectancy of less than 72 hours.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The participates had received their first orthotopic liver transplantation within 10 days prior. And there are no gender restrictions. The number of participants are 800.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Clinically significant CMV reactivation or CMV disease was observed within 12 months of transplantation | Within 22 months after liver transplantation
  1. CMV reactivation: CMV-lgG is positive and any one of CMV-lgM, pp65 and CMV-DNA is positive is called CMV reactivation.
End of follow-up survey | Within 22 months after liver transplantation
  We will perform a follow-up for 22 months if participant is alive and does not observed CMV reactivation.
Death | Within 22 months after liver transplantation
  The participant died

SECONDARY OUTCOMES:
Loss to follow-up survey | Within 22 months after liver transplantation
  During follow-up, if we can not connect with participant, we regard this event as loss to follow-up.
Participants asked to withdraw | Within 22 months after liver transplantation
  During follow-up, participants refuse to keep this study within 22 months after liver transplantation

IPD SHARING:
Plan to Share IPD: Undecided